CLINICAL TRIAL: NCT07009379
Title: Pillow Brace Assessment on Sleep Quality of Patients Undergoing Arthroscopic Rotator Cuff Surgery
Acronym: PILLOW BRACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-A00036-43
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Rotator Cuff Injury
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pillow Brace (Experimental): The "Pillow Brace" arm will consist of a Dujarrier-type splint to which a deformable cushion will be fixed
  Interventions: Device: Intervention A
- Standard (Other): The "Standard" arm will consist of a Dujarrier-type splint
  Interventions: Device: Intervention B

INTERVENTIONS:
Device: Intervention A — Intervention A means Pillow Brace
  Arms: Pillow Brace
Device: Intervention B — Intervention B means standard management
  Arms: Standard

SUMMARY:
Rotator cuff surgery is an increasingly popular procedure in France. It is a common procedure for patients with shoulder tendon injuries, aimed at restoring mobility and reducing pain. Although arthroscopic techniques have improved functional outcomes, managing postoperative pain, particularly at night, and its consequences remains a major challenge.

Studies highlight that postoperative nighttime pain can significantly affect sleep quality, delaying functional recovery and patient satisfaction. However, standard splints used for postoperative immobilization do not offer an optimal solution to this problem, leaving a significant gap in the care of these patients.

Given this observation, a splint incorporating a support cushion system could meet the specific needs expressed by patients who have undergone rotator cuff surgery, namely improving sleep quality by minimizing nighttime pain. This splint, called the "Pillow Brace," was developed internally at the Jouvenet Clinic. It therefore does not have CE marking.

Nevertheless, this study is based on the hypothesis that the use of a "Pillow Brace" could significantly improve sleep quality compared to standard splints, thus making a significant contribution to orthopedic medicine, postoperative rehabilitation, and patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing arthroscopic rotator cuff repair surgery confirmed by clinical diagnosis and preoperative imaging tests.
* Patient able to understand the instructions for using the brace.
* Patient able to perform activities of daily living with or without a brace, ensuring proper use of the brace.
* Patient affiliated with or beneficiary of a social security system
* French speaking patient, having signed an informed consent form

Exclusion Criteria:

* Patient with an uncertain diagnosis
* Patient undergoing rotator cuff revision surgery.
* Patient with complex or surgical fractures of the shoulder, humerus, or ribs
* Patient with multiple fractures, open fractures, or those with pinning
* Patient who has undergone multiple surgeries in the last 6 months.
* Patient with shoulder pathologies unrelated to the rotator cuff, such as severe arthritis or capsulitis.
* Patient on long-term morphine treatment
* Patient with known allergies to splint materials
* Protected patient: adult under guardianship, curatorship, or other legal protection, deprived of liberty by judicial or administrative order
* Pregnant woman
* Patient hospitalized without consent
* Patient already enrolled and participating in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | Month 1
  Sleep quality will be assessed using PSQI (Pittsburg Sleep Qulity Index). Score is from 0 to 21. 0 means no sleel problems whereas 21 means major sleep problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Jouvenet, Paris, France